CLINICAL TRIAL: NCT03027531
Title: eKISS Electronic KIOSK Intervention for Safer-Sex: A Pilot Randomized Controlled Trial of an Interactive Computer-based Intervention for Sexual Health in Adolescents and Young Adults
Brief Title: eKISS: Electronic KIOSK Intervention for Safer-Sex
Acronym: eKISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Taraneh Shafii, Associate Professor, Department of Pediatrics, Division of Adolescent Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 32030-B; 5K23HD052621 (NIH)
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Reproductive Behavior; Contraception; Sexually Transmitted Diseases
Keywords: reproductive health, condoms, sexually transmitted diseases, contraception
MeSH Terms: conditions — Reproductive Behavior; Sexually Transmitted Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Control group entered sexual history via computer assisted self-interview and provided specimens for chlamydia, gonorrhea and pregnancy(females) testing. The do not receive the feedback intervention of eKISS: electronic KIOSK for safer-sex
  Interventions: Behavioral: eKISS: electronic KIOSK for Safer-Sex
- Intervention (Experimental): Intervention group entered sexual history via computer assisted self-interview and received the interactive computer-based intervention with individualized feedback eKISS: electronic KIOSK for safer-sex. They provided specimens for chlamydia, gonorrhea and pregnancy(females) testing.
  Interventions: Behavioral: eKISS: electronic KIOSK for Safer-Sex

INTERVENTIONS:
Behavioral: eKISS: electronic KIOSK for Safer-Sex — An interactive computer-based intervention for safer-sex which provides individualized feedback about protective and risky sexual behaviors; offers instructive video modules for safe-sex; elicits change behavior and identification of behavior change goal using elements of motivational interviewing.

SUMMARY:
This study is a randomized controlled trial to test acceptability, feasibility and preliminary efficacy of an interactive computer-based intervention with individualized feedback to promote sexual health in adolescents and young adults with assessment of behavioral and biomarker outcomes.

DETAILED DESCRIPTION:
This study is a randomized controlled trial to test acceptability, feasibility and preliminary efficacy of an interactive computer-based intervention (ICBI) with individualized feedback to promote sexual health in adolescents and young adults. The intervention uses physician avatars and uses elements of motivational interviewing to elicit sexual risk behaviors and motivation to change risky behavior. Feedback includes instructive video modules. Participants were asked to identify one behavior to change and were reassessed at 3-month follow-up for interim sexual behavior including condom and birth control use. Participants were tested for chlamydia, gonorrhea, and pregnancy(females) at baseline and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* English speaking and reading
* Report at least one episode of unprotected vaginal sex (no condom OR no birth control) in the last 2 months
* Not currently pregnant or actively seeking pregnancy in self or partner

Exclusion Criteria:

* Currently pregnant or actively seeking pregnancy in self or partner

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 272 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Unprotected sex (no condoms) from self-report via computerized survey | during last 2 months (asked at 3 month follow-up visit)
  number of unprotected sex events when participant did not use condom during sex

SECONDARY OUTCOMES:
Unprotected sex (no birth control) from self-report via computerized survey | during last 2 months (asked at the 3-month follow-up visit)
  number of unprotected sex events when participant did not use birth control during sex
Number of sex partners from self-report via computerized survey | during last 2 months (asked at the 3-month follow-up visit)
  number of partners with which the participant had sex
Biomarkers: urine sample tested with nucleic acid amplification test for STDs and urine sample pregnancy test | over last 3 months (asked at the 3-month follow-up visit)
  Incident chlamydia, gonorrhea, and pregnancy since baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Taraneh Shafii, MD, MPH, Principal Investigator — University of Washington; King K Holmes, MD, PhD, Principal Investigator — University of Washington; Center for AIDS and STD

IPD SHARING:
Plan to Share IPD: No